CLINICAL TRIAL: NCT01850030
Title: A Double-Blind, Double-Dummy, Randomized, Two-arm, Multicenter Study Comparing the Efficacy, Safety and Tolerability of Oral Dydrogesterone 30 mg Daily Versus Intravaginal Micronized Progesterone Capsules 600 mg Daily for Luteal Support in In-Vitro Fertilization (Lotus I)
Brief Title: A Multicenter Study Comparing the Efficacy, Safety and Tolerability of Oral Dydrogesterone 30 mg Daily Versus Intravaginal Micronized Progesterone Capsules 600 mg Daily for Luteal Support in In-Vitro Fertilization
Acronym: Lotus I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-563; 2012-002215-26 (EudraCT Number)
Record Dates: First submitted 2013-04-19; First posted 2013-05-09 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-05

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Dydrogesterone; Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dydrogesterone 30 mg (Experimental)
  Interventions: Drug: Dydrogesterone 30 mg; Drug: Placebo progesterone
- Micronized Progesterone 600 mg (Experimental)
  Interventions: Drug: Micronized Progesterone 600 mg; Drug: Placebo dydrogesterone

INTERVENTIONS:
Drug: Dydrogesterone 30 mg — Oral Dydrogesterone 10 mg tablets tid
  Arms: Dydrogesterone 30 mg
Drug: Micronized Progesterone 600 mg — Intravaginal micronized progesterone 200 mg capsules tid
  Arms: Micronized Progesterone 600 mg
Drug: Placebo progesterone — Placebo intravaginal micronized progesterone 200 mg capsules tid
  Arms: Dydrogesterone 30 mg
Drug: Placebo dydrogesterone — placebo oral dydrogesterone 10 mg tablets tid
  Arms: Micronized Progesterone 600 mg

SUMMARY:
Female inability to conceive a child. The purpose of this randomized, two-arm and double blind, double dummy study is to demonstrate that the treatment of a daily dose of 3x10mg dydrogesterone orally is as effective and safe as the daily dose of 3x200 mg micronized progesterone capsules administered intravaginally for the luteal support in patients undergoing IVF. The treatment will start on the day of oocyte retrieval and continue until pregnancy is negative or until week 12 gestation.Patients will be followed after treatment until 30 days after delivery to record any safety and tolerability data of the patient and their newborn(s).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Premenopausal females, age > 18 years < 42 years
* Non-smokers. For females who were past smokers, they must have stopped tobacco usage for at least 3 months prior baseline visit
* Early follicular phase (Day 2-4) Follicle stimulating hormone (FSH) less than or equal to 15 IU/L and estradiol (E2)within normal limits
* Luteinizing hormone (LH), prolactin (PRL), T (testosterone) and thyroid-stimulating hormone (TSH), within the normal limits for the clinical laboratory, or considered not clinically significant by the Investigator within 6 months prior to screening
* Documented history of infertility (e.g., unable to conceive for at least one year or for 6 months for women ≥ 38 years of age or bilateral tubal occlusion or absence)
* Normal transvaginal ultrasound at screening (or within 14 days of screening) without evidence of clinically significant abnormality consistent with finding adequate for Assisted Reproductive Technology (ART) with respect to uterus and adnexa (no hydrosalpinx or clinically relevant uterine fibroids)
* Negative pregnancy test on the day of pituitary down regulation (prior to administration of gonadotropin releasing hormones (GnRH) agonist or GnRH antagonist)
* Clinically indicated protocol for induction of IVF with a fresh embryo
* Single or dual embryo transfer
* BMI ≥ 18 and ≤ 30 kg/m2

Exclusion Criteria:

* Evidence of cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematologic/immunologic, head, ears, eyes, nose, throat (HEENT), dermatologic/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurologic/psychiatric, allergy, recent major surgery (< 3 months), or other relevant diseases as revealed by history, physical examination and/or laboratory assessments which could limit participation in or completion of the study
* Acute urogenital disease
* Known allergic reactions to progesterone products
* Known allergic reactions to peanuts and peanut oil
* Intake of experimental drug or participation in any other clinical trial within 30 days prior to study start
* Mental disability or any other lack of fitness, in the Investigator's opinion, to preclude subjects to participate in or to complete the study
* Current or recent substance abuse, including alcohol and tobacco (Note: Patients who stopped tobacco usage at least 3 months prior to screening visit would be allowed)
* History of chemotherapy or radiotherapy
* Patients with more than 3 unsuccessful IVF attempts
* Contraindication for pregnancy
* Refusal or inability to comply with the requirements of the study protocol for any reason, including scheduled clinic visits and laboratory tests
* History of recurrent pregnancy loss defined as 3 or more spontaneous miscarriages

Ages: 19 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1070 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darline Cheatham-Seitz, MD, PhD, Study Director — Abbott
Locations (39):
- Site reference no. 113176, Vienna, Austria
- Belgium (10):
  - Site reference no. 93593, Brasschaat
  - Site reference no. 93598, Brussels
  - Site reference no. 93615, Brussels
  - Site reference no. 93617, Brussels
  - Site reference no. 93613, Genk
  - Site reference no. 93594, Ghent
  - Site reference no. 93597, Ghent
  - Site reference no. 93616, Hasselt
  - Site reference no. 93595, Leuven
  - Site reference no. 93614, Mons
- Finland (5):
  - Site reference ID ORG-000884, Helsinki
  - Site reference ID ORG-000885, Jyväskylä
  - Site reference no. ORG-000635, Oulu
  - Site reference ID ORG-000795, Tampere
  - Site reference no. ORG-000633, Turku
- Germany (5):
  - Site reference ID ORG-000645, Berlin
  - Site reference ID ORG-000643, Berlin
  - Site reference ID ORG-000642, Dresden
  - Site reference ID ORG-000644, Heidelberg
  - Site reference ID ORG-000883, Lübeck
- Israel (5):
  - Site reference no. 93635, Beersheba
  - Research facility ID ORG-000934, Hadera
  - Research facility ID ORG-000935, Haifa
  - Site reference no. 93638, Jerusalem
  - Site reference no. 93641, Tel Aviv
- Russia (7):
  - FGBU Endocrinology Research Center of Minzdrav of Russia, Moscow
  - Moscow State Medical Dentistry University, Moscow
  - CJSC "Nasledniki", Moscow
  - SBEIHPE - NWSMU n.a.l.l.Melnichko MoH and SD of RF, Saint Petersburg
  - St. Petersburg SBHI "Maternity Hospital No 17" (main address), Saint Petersburg
  - FSBI "Ural SRI of Maternity and Child Protection" of MoH and SD, Yekaterinburg
  - Center of Family Medicine LC, Yekaterinburg
- Spain (6):
  - Site reference no. 119915, Baracaldo, Vizcaya
  - Site reference ID ORG-000791, Barcelona
  - Site reference no. ORG-000639, Bilbao
  - Site reference no. ORG-000640, Pozuelo de Alarcon (Madrid)
  - Site reference no. ORG-000638, Seville
  - Site reference no. ORG-000637, Valencia

REFERENCES:
- [Derived] Tournaye H, Sukhikh GT, Kahler E, Griesinger G. A Phase III randomized controlled trial comparing the efficacy, safety and tolerability of oral dydrogesterone versus micronized vaginal progesterone for luteal support in in vitro fertilization. Hum Reprod. 2017 May 1;32(5):1019-1027. doi: 10.1093/humrep/dex023. PMID 28333318

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1070 subjects were enrolled in the study and 1031 subjects were randomized
Period: Overall Study
Arm/Group | Dydrogesterone 30 mg | Micronized Progesterone 600 mg
Started | 520 | 511
Completed | 173 | 142
Not Completed | 347 | 369
Not completed — Adverse Event | 64 | 82
Not completed — Lack of Efficacy | 3 | 1
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 24 | 28
Not completed — pregnancy not confirmed at visit 4 | 248 | 249

BASELINE CHARACTERISTICS:
Population: The full analysis sample was used here which consists of all subjects that received at least one administration of study drug and had a successful embryo transfer performed at Visit 3 (Day 3 to 6) or did not prematurely discontinue prior to embryo transfer at Visit 3 (Day 3 to 6) due to non-study drug-related issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dydrogesterone 30 mg | Micronized Progesterone 600 mg | Total
Number analyzed (Participants) | 497 | 477 | 974
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 497 | 477 | 974
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (4.5) | 32.5 (4.4) | 32.5 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 497 | 477 | 974
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 7 | 7 | 14
  Russian Federation | 106 | 103 | 209
  Belgium | 194 | 182 | 376
  Finland | 4 | 5 | 9
  Israel | 69 | 66 | 135
  Germany | 62 | 60 | 122
  Spain | 55 | 54 | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Being Pregnant as Measured by the Presence of Fetal Heart Beats at 12 Weeks´Gestation Using Transvaginal Ultrasound
Description: Percentage of participants being pregnant as measured by the presence of fetal heart beats at 12 weeks´gestation using transvaginal ultrasound
Time Frame: 12 weeks´ gestation (at visit 6)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dydrogesterone 30 mg | Micronized Progesterone 600 mg
Number analyzed (Participants) | 497 | 477
percentage of participants | 37.6 [33.4 to 42.1] | 33.1 [28.9 to 37.6]

2. Secondary Outcome: Percentage of Participants Being Pregnant as Measured by the Positive Biochemical Pregnancy Test on Day 14 After Embryo Transfer
Description: Percentage of participants being pregnant as measured by the positive biochemical pregnancy test on Day 14 after embryo transfer
Time Frame: Day 14 after embryo transfer
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dydrogesterone 30 mg | Micronized Progesterone 600 mg
Number analyzed (Participants) | 497 | 477
percentage of participants | 47.1 [42.6 to 51.6] | 45.5 [41.0 to 50.1]

3. Secondary Outcome: Percentage of Participants With a Successful Completion of Pregnancy
Description: Incidence of live births and healthy newborns
Time Frame: After delivery (about 9 months after IVF)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dydrogesterone 30 mg | Micronized Progesterone 600 mg
Number analyzed (Participants) | 497 | 477
percentage of participants
  Live birth rate | 34.6 [30.4 to 39.0] | 29.8 [25.7 to 34.1]
  Healthy newborn rate | 32 [27.9 to 36.3] | 27.7 [23.7 to 31.9]

4. Secondary Outcome: Gender of the Newborn
Description: was recorded and collected for Newborn
Time Frame: After delivery (about 9 months after IVF)
Measure: Number; unit: number of newborns
Arm/Group | Dydrogesterone 30 mg | Micronized Progesterone 600 mg
Number analyzed (Participants) | 213 | 158
number of newborns
  Gender male | 120 | 88
  Gender female | 93 | 70

ADVERSE EVENTS:
Description: For Adverse Events reporting the safety sample was used consisting of all subjects which have received at least one administration of study drug (518 subjects in Dydrogesterone, 511 subjects in Micronized Progesterone)
Arm/Group | Dydrogesterone 30 mg | Micronized Progesterone 600 mg
Serious Adverse Events (participants affected / at risk) | 56/518 | 68/511
Other Adverse Events (participants affected / at risk) | 156/518 | 147/511
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dydrogesterone 30 mg (N=518) | Micronized Progesterone 600 mg (N=511)
spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 16 (16)
abortion not specified as induced or spontaneous (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 11 (11)
maternal complications of pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 7 (7)
labor onset and length abnormalities (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 5 (7)
Still birth and foetal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 6 (6)
Foetal complications NEC (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3)
Hypertension associated disorders of pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (3) | 2 (3)
Amniotic fluid and cavity disorders of pregnancy NEC (Pregnancy, puerperium and perinatal conditions) | 2 (3) | 1 (1)
Gestational age and weight conditions (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Haemorrhagic complications of pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (3)
High risk pregnancies (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Normal pregnancy, labour and delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Umbilical cord complications (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Abortion related conditions and complications (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
foetal growth complications (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
maternal complications of delivery NEC (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Postpartum complications NEC (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ovarian and fallopian tube disorders NEC (Reproductive system and breast disorders) | 8 (8) | 6 (7)
Cervix disorders (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Ovarian and fallopian tube cysts and neoplasms (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Menstruation and uterine bleeding NEC (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive tract disorders NEC (excl neoplasms) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal disorders NEC (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Induced abortions (Surgical and medical procedures) | 3 (3) | 4 (4)
Obstetric therapeutic procedures (Surgical and medical procedures) | 1 (1) | 0 (0)
Autosomal chromosomal abnormalities (Congenital, familial and genetic disorders) | 1 (1) | 3 (3)
Arterial disorders congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cardiac septal defects congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cardiac valve disorders congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Central nervous system disorders congenital NEC (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cerebral disorders congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Sex chromosomal abnormalities (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Gastrointestinal and abdominal pains (excl oral and throat) (Gastrointestinal disorders) | 1 (1) | 4 (4)
Peripheral embolism and thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Vascular hypertensive disorders NEC (Vascular disorders) | 1 (2) | 1 (1)
haemorrhages NEC (Vascular disorders) | 0 (0) | 1 (1)
Abdominal and gastrointestinal infections (Infections and infestations) | 0 (0) | 1 (1)
cytomegaloviral infections (Infections and infestations) | 0 (0) | 1 (1)
infections NEC (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infections (Infections and infestations) | 0 (0) | 1 (1)
non-site specific injuries NEC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal and urinary tract injuries NEC (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Autonomic nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1)
Neurological signs and symptoms NEC (Nervous system disorders) | 1 (1) | 0 (0)
Seizures and seizure disorders NEC (Nervous system disorders) | 1 (1) | 0 (0)
Rate and rythm disorders NEC (Cardiac disorders) | 1 (1) | 1 (1)
Foetal and neonatal diagnostic procedures (Investigations) | 1 (1) | 0 (0)
protein analyses NEC (Investigations) | 0 (0) | 1 (1)
Anaemias NEC (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenias (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Potassium imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Urinary abnormalities (Renal and urinary disorders) | 1 (1) | 0 (0)
Nasal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dydrogesterone 30 mg (N=518) | Micronized Progesterone 600 mg (N=511)
Vaginal haemorrhage (Reproductive system and breast disorders) | 61 (75) | 45 (53)
Procedural pain (Injury, poisoning and procedural complications) | 38 (39) | 41 (42)
Nausea (Gastrointestinal disorders) | 44 (46) | 26 (27)
Abdominal pain (Gastrointestinal disorders) | 24 (25) | 31 (33)
Headache (Nervous system disorders) | 27 (31) | 32 (36)
Pregnancy of unknown location (Pregnancy, puerperium and perinatal conditions) | 19 (19) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the Site shall provide to Sponsor a copy of all such manuscripts and materials, and allow sponsor sixty (60) days to review and comment on them.

If the Sponsor requests, the Site shall remove any Confidential Information (other than Study results) prior to submitting or presenting the materials.